CLINICAL TRIAL: NCT00000113
Title: Correction of Myopia Evaluation Trial (COMET)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NEI-9; U10EY011756 (NIH)
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Myopia
Keywords: myopia; nearsightedness
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progressive Addition Lenses (PALs) (Experimental)
  Interventions: Other: Progressive Addition Lenses
- Single Vision Lenses (Active Comparator)
  Interventions: Other: single vision lenses

INTERVENTIONS:
Other: Progressive Addition Lenses — Varilux comfort with +2.00 addition
  Arms: Progressive Addition Lenses (PALs)
Other: single vision lenses
  Arms: Single Vision Lenses

SUMMARY:
To evaluate whether progressive addition lenses (PALs) slow the rate of progression of juvenile-onset myopia (nearsightedness) when compared with single vision lenses, as measured by cycloplegic autorefraction. An additional outcome measure is axial length, as measured by A-scan ultrasonography.

To describe the natural history of juvenile-onset myopia in a group of children receiving conventional treatment (single vision lenses).

DETAILED DESCRIPTION:
Myopia (nearsightedness) is an important public health problem, which entails substantial societal and personal costs. It is highly prevalent in our society and even more frequent in Asian countries; furthermore, its prevalence may be increasing over time. High myopia contributes to significant loss of vision and blindness. At present, the mechanisms involved in the etiology of myopia are unclear, and there is no way to prevent the condition. Current methods of correction require lifelong use of lenses or surgical treatment, which is expensive and may lead to complications. The rationale for this trial, the Correction of Myopia Evaluation Trial (COMET), arises from the convergence of research involving (1) the link between accommodation and myopia in children and (2) animal models of myopia showing the important role of the visual environment in eye growth. A contribution of this research is that blur is a critical component in the development of myopia. The primary aim of COMET, to evaluate the efficacy of progressive addition lenses, a noninvasive intervention, in slowing the progression of myopia, follows from this line of reasoning. These lenses should provide clear visual input over a range of viewing distances without focusing effort by the child. The comparison of myopia progression in children treated with PALs versus single vision lenses will allow the quantification of the effect of PALs on myopia progression during the followup period.

The COMET is a multicenter, randomized, double-masked clinical trial to evaluate whether PALs slow the progression of juvenile-onset myopia as compared with single vision lenses. The study is a collaborative effort that involves a Study Chair at the New England College of Optometry; four clinical centers at colleges of optometry in Boston, Birmingham, Philadelphia, and Houston; and a Coordinating Center at the State University of New York at Stony Brook.

The sample size goal, 450 children with myopia in both eyes who met specific inclusion and exclusion criteria, was attained with the enrollment of 469 children in one year. Children were identified from school screenings, clinic records, and referrals from local practitioners. Eligible children were randomly assigned to receive progressive addition or single vision lenses. Participating children are being examined at 6-month intervals following baseline, for at least 3 years, to measure changes in refractive error and to update prescriptions, according to a specified protocol. A dilated examination to evaluate the study outcome measures is performed at the annual study visits. A standardized, common protocol is used at all centers.

The primary outcome of the study is progression of myopia, defined as the magnitude of the change relative to baseline in spherical equivalent refraction, determined by cycloplegic autorefraction. The secondary outcome of the study is axial length measured by A-scan ultrasonography.

ELIGIBILITY:
Children between the ages of 6 and 12 years with myopia in both eyes (defined as spherical equivalent between -1.25 D and -4.50 D in each eye as measured by cycloplegic autorefraction), astigmatism less than or equal to 1.50 D, and no anisometropia (defined as a difference in spherical equivalent between the two eyes greater than 1.0 D) are eligible for inclusion. Exclusion criteria include visual acuity greater than 20/25, strabismus, use of contact lenses, birth weight less than 1,250 grams, use of bifocal or progressive addition lenses, or any conditions precluding adherence to the protocol.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 469 (Actual)
Dates: Start 1997-09; Primary Completion 2001-10 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Progression of myopia, determined by cycloplegic autorefraction

SECONDARY OUTCOMES:
Axial length measured by A-scan ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Jane Gwiazda, PhD, Study Chair — New England College of Optometry; Leslie Hyman, PhD, Study Director — Stony Brook Medicine
Locations (4):
- United States (4):
  - University of Alabama-Birmingham, School of Optometry, Birmingham, Alabama
  - New England College of Optometry, Boston, Massachusetts
  - Pennsylvania College of Optometry, Philadelphia, Pennsylvania
  - University of Houston, College of Optometry, Houston, Texas

REFERENCES:
- [Result] Gwiazda J, Hyman L, Hussein M, Everett D, Norton TT, Kurtz D, Leske MC, Manny R, Marsh-Tootle W, Scheiman M. A randomized clinical trial of progressive addition lenses versus single vision lenses on the progression of myopia in children. Invest Ophthalmol Vis Sci. 2003 Apr;44(4):1492-500. doi: 10.1167/iovs.02-0816. PMID 12657584
- [Result] Gwiazda JE, Hyman L, Norton TT, Hussein ME, Marsh-Tootle W, Manny R, Wang Y, Everett D; COMET Grouup. Accommodation and related risk factors associated with myopia progression and their interaction with treatment in COMET children. Invest Ophthalmol Vis Sci. 2004 Jul;45(7):2143-51. doi: 10.1167/iovs.03-1306. PMID 15223788
- [Result] Hyman L, Gwiazda J, Hussein M, Norton TT, Wang Y, Marsh-Tootle W, Everett D. Relationship of age, sex, and ethnicity with myopia progression and axial elongation in the correction of myopia evaluation trial. Arch Ophthalmol. 2005 Jul;123(7):977-87. doi: 10.1001/archopht.123.7.977. PMID 16009841
- [Derived] Lawrenson JG, Shah R, Huntjens B, Downie LE, Virgili G, Dhakal R, Verkicharla PK, Li D, Mavi S, Kernohan A, Li T, Walline JJ. Interventions for myopia control in children: a living systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 16;2(2):CD014758. doi: 10.1002/14651858.CD014758.pub2. PMID 36809645
- [Derived] Deng L, Gwiazda J, Manny RE, Scheiman M, Weissberg E, Fern KD, Weise K; COMET Study Group. Limited change in anisometropia and aniso-axial length over 13 years in myopic children enrolled in the Correction of Myopia Evaluation Trial. Invest Ophthalmol Vis Sci. 2014 Apr 3;55(4):2097-105. doi: 10.1167/iovs.13-13675. PMID 24576881
- [Derived] Gwiazda J, Deng L, Manny R, Norton TT; COMET Study Group. Seasonal variations in the progression of myopia in children enrolled in the correction of myopia evaluation trial. Invest Ophthalmol Vis Sci. 2014 Feb 4;55(2):752-8. doi: 10.1167/iovs.13-13029. PMID 24408976